CLINICAL TRIAL: NCT02609815
Title: Effect of INitial Combination Therapy With GEmigliptin and Metformin on Microbiota Change and Glycemic Control in patientS With Type 2 DIabetes aNd ObEsity (INTESTINE Study)
Brief Title: Initial Combination of Gemigliptin and Metformin on Microbiota Change
Acronym: INTESTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-INTESTINE2015
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — LC15-0444; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemigliptin/metformin (Experimental): zemimet-SR 50/1000 mg x 1 tablet
  Interventions: Drug: gemigliptin/metformin
- glimepiride/metformin (Active Comparator): amaryl-Mex 1/500 mg x 2 tablets
  Interventions: Drug: glimepiride/metformin

INTERVENTIONS:
Drug: gemigliptin/metformin — zemimet-SR 50/1000 mg x 1 tablet
  Other Names: Zemimet
  Arms: gemigliptin/metformin
Drug: glimepiride/metformin — amaryl-Mex 1/500 mg x 2 tablets
  Other Names: Amarylmex
  Arms: glimepiride/metformin

SUMMARY:
The purpose of this study is to investigate gut microbiota change and glucose lowering effect of initial combination therapy of gemigliptin and metformin compared to glimepiride and metformin in obese patients with type 2 diabetes.

DETAILED DESCRIPTION:
Obese type 2 diabetes patients who were not treated with anti-diabetic medication within 6 weeks, were randomly assigned to gemigliptin/metformin or sulphonylurea/metformin. After 24 week treatment, gut microbiota composition change, glucose lowering effect, body weight, and gut hormones were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Drug naive (no anti-diabetic medication within 6 weeks)
* HbA1c >= 7.5%
* BMI >= 25.0 kg/m2

Exclusion Criteria:

* Type 1 diabetes
* DKA, HHS
* history of hypersensitivity to sulphonylurea, metformin or DPP-4 inhibitor
* Gestational diabetes mellitus
* Serum Cr >1.5 mg/dL (male), >1.4mg/dL (female)
* Abnormal liver function test
* Anti-obesity medication within 3 months
* Gastrointestinal motility drug, laxatives within 3 months
* History of major gastrointestinal surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
gut microbiota composition change from baseline | 24 weeks
  Analysis of gut microbiota composition at class, genus, and species levels before and after treatment. Inter-individual changes of gut microbiota changes were analyzed.

SECONDARY OUTCOMES:
HbA1c change | 24 weeks
  HbA1c change from baseline to 24 weeks

OTHER OUTCOMES:
Body composition | 24 weeks
  Using bioimpedance analysis, muscle mass and total and visceral fat mass were analyzed after 24 week treatment.
Beta-cell function | 24 weeks
  HOMA-beta and insulinogenic index calculated before and after treatment.
GLP-1 | 24 weeks
  Plasma levels of GLP-1 during 75g OGTT.
GIP | 24 weeks
  Plasma levels of GIP during 75g OGTT.
PYY | 24 weeks
  Plasma levels of PYY during 75g OGTT.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Jung Oh, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No